CLINICAL TRIAL: NCT03850847
Title: Understanding Decision Making in the Intensive Care Unit: a National Study
Status: Active, not recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CE 18.323
Record Dates: First submitted 2019-02-15; First posted 2019-02-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Organ Donation
Keywords: Neurological Determination of Death; Organ Donation; Determination of Death; Understanding Decision Making; Substitute Decision Maker
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multi-Methods Study: Step 1: Semi-structured Interviews
  Step 2: National Telephone Survey
  Interventions: Other: Step 1: Semi-structured Interviews; Other: Step 2: National Telephone Survey

INTERVENTIONS:
Other: Step 1: Semi-structured Interviews — 1. Cover SDMs' experience around:
     * withdrawal of life sustaining therapies
     * organ donation among those who were approached (including with the medical team and the organ donation organisation)
     * understanding of the situation
     * views on any gaps in the quantity or quality of information and discussion they received concerning their loved one's end-of-life care or donation process
  2. Explore factors they perceived to influence their decision to consent to organ donation or not (or that would have influenced their decision for those not approached), and how such factors may have changed over the course of making this decision and since the decision (or since the event for those not approached).
Other: Step 2: National Telephone Survey — Explore SDM's beliefs and experiences around end of life and assess which beliefs are associated with the decision taken at the end of life, including decision to donate organs or not (and the strength of this association)

SUMMARY:
Given how central Substitute Decision Makers (SDMs) are to the process leading to end of life decisions and sometimes, organ donation, it is striking how poorly understood this decision-making process is. A 2017 scoping review on the topic of soliciting SDM consent to organ donation reported on more than 168 studies covering a broad range of topics, including: SDM characteristics and predictors of consent; the process of soliciting consent; and the effect of the decision on subsequent process of care and on family well-being. An unexplored area, however, is factors - including modifiable factors - that influence SDM decision making at the end of life, which organ donation is part of, such as: responses to stress, support from extended families and friends, and personal beliefs about the ongoing medical conditions. This project seeks to fill this clear and important gap.

In the ICU, at the end of life, SDMs are under incredible emotional distress, have often not eaten or slept properly for days preceding discussions about end of life and organ donation, and are also in the midst of grieving for their loved one. The time pressure poses challenges for SDMs' decision making. Thus, this study will investigate novel, potentially modifiable reasons for end of life decision so that we may better support this personally challenging and important decision, especially if organ donation decision interferes with the decision process.

Primary objective: To investigate beliefs and experiences of SDMs involved in the decision-making process around withdrawal of life sustaining therapies .

Secondary objective: To inform efforts to improve support for SDMs with the aim of improving the decision-making process end-of-life decisions, including when organ donation is involved.

DETAILED DESCRIPTION:
A national multicenter multi-methods study with SDMs will be conducted in two steps. In Step 1, a semi-structured interviews with SDMs will be conducted. The sampling frame will balance interviews with those that were approached or not for organ donation, and consented or not to organ donation. Interviews will be informed by two complementary theoretical frameworks. Building on Step 1 results, in Step 2 a national telephone survey of SDMs will be conducted to test which factors are associated with end-of-life decisions.

ELIGIBILITY:
Inclusion Criteria:

* Substitute decision maker (SDM) and patients with at least 18 years old
* SDM(s) of patients in the ICU with or without brain injury for whom withdrawal of life-sustaining therapies is considered or has been discussed.
* SDM(s) of patients for whom death is expected to occur within approximately 1 hour after withdrawal of life-sustaining therapies
* English or French speakers SDM(s)
* SDM(s) reachable in ICU

Exclusion Criteria:

* SDM is not reachable after pre-consent in ICU (after 5 initial attempts within a 3-week period).
* SDM asks to postpone the interview more than 3 times.
* SDM unable to provide informed verbal consent for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surogate decision makers of critically ill deceased patients, potential organ donors. Are included all SDMs, whether the patient donated organs or not, or were approached for organ donation or not, thus providing a global view of the decision making at the end of life and how it is affected by organ donation, or how it affects organ donation when appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
SDM's beliefs and experiences around end of life | 6 weeks to 2 months after patient's hospitalisation in the intensive care unit
  Assess which beliefs and experiences are associated with the decision to donate organs using open-ended questions. The responses obtained from the interviews will be analysed and classified based on the Leventhal's Common Sense Self-Regulation Model and the theoretical domain Framework. The most significant domains will help inform the creation of a larger scale national survey to help investigate what domains affect decision-making around end of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chassé, MD PhD FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (9):
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crawshaw J, Presseau J, van Allen Z, Pinheiro Carvalho L, Jordison K, English S, Fergusson DA, Lauzier F, Turgeon AF, Sarti AJ, Martin C, D'Aragon F, Li AH, Knoll G, Ball I, Brehaut J, Burns KEA, Fortin MC, Weiss M, Meade M, Marsolais P, Shemie S, Zaabat S, Dhanani S, Kitto SC, Chasse M; Canadian Donation and Transplantation Research Program and the Canadian Critical Care Trials Group. Exploring the experiences and perspectives of substitute decision-makers involved in decisions about deceased organ donation: a qualitative study protocol. BMJ Open. 2019 Dec 23;9(12):e034594. doi: 10.1136/bmjopen-2019-034594. PMID 31874899